CLINICAL TRIAL: NCT07076446
Title: An Open-label, Multicenter Study to Assess the Pharmacokinetics, Safety, and Tolerability of Immune Globulin Subcutaneous (Human) IgPro20 in IG Treatment-naïve Subjects With Primary Immunodeficiency
Brief Title: An Open-label, Multicenter Study to Assess the Pharmacokinetics (PK), Safety, and Tolerability of Subcutaneous IgPro20 in Immunoglobulin (IG) Treatment-naïve Participants With Primary Immunodeficiency (PID)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IgPro20_4007
Record Dates: First submitted 2025-07-15; First posted 2025-07-22 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-07

CONDITIONS: Primary Immunodeficiency
Keywords: Immunoglobulin replacement therapy
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — gamma-Globulins; Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IgPro20 (Experimental): All participants will receive a loading dose of IgPro20 daily from Day 1 to 5 in Week 1, followed by weekly administration of the maintenance dose of IgPro20 from Day 8 (Week 2) to Day 78 (Week 12).
  Interventions: Biological: IgPro

INTERVENTIONS:
Biological: IgPro — IgPro20 is a solution for infusion for subcutaneous administration.
  Other Names: Immune globulin subcutaneous (Human) 20% liquid

SUMMARY:
This is an open-label, multicenter, phase 4 study in IG treatment-naïve participants with PID, conducted in the United States (US), to assess the PK, safety, and tolerability of IgPro20. The primary objective of this study is to characterize the PK of IgPro20 and to assess the safety and tolerability of IgPro20 in IG treatment-naïve participants with PID who are aged greater than or equal to (>=) 18 years.

ELIGIBILITY:
Inclusion Criteria:

* - Participants must be aged >=18 years.
* - Participants must have a confirmed and documented diagnosis of PID, must be IG treatment-naïve and have an IgG level less than or equal to (<=) 400 milligrams per deciliter(mg/dL) at Screening.

Exclusion Criteria:

* - Participants with hyperprolinemia.
* - Participants who are receiving the following medications:
* • Systemic corticosteroids (prednisone or equivalent; average daily dose of greater than [>] 15 mg) from 4 weeks before Screening.
* • Any dose of systemic immunosuppressants within 9 months or 5 times the half-life (t½) plus 6 months before Screening, whichever is longer.
* • Any dose of biologic therapies with influence on the immune system (eg, tumor necrosis factor inhibitors, interleukin inhibitors, B-cell inhibitors), including investigational agents, within 12 months or 5 times the t½ plus 6 months before Screening, whichever is longer.
* • Participants who are currently receiving anti-coagulation therapy.
* - Participants with hypoalbuminemia, protein-losing enteropathies, and kidney diseases with proteinuria.
* - Participants with a documented history or a current diagnosis of a thromboembolic event(s) (eg, deep vein thrombosis, pulmonary embolism, myocardial infarction, cerebrovascular accident, transient ischemic attack) or coagulopathy within 12 months before Screening.
* - Participants with severe dehydration and known blood disorders affecting viscosity.
* - Participants with aspartate aminotransferase and alanine aminotransferase concentration > 3 times the upper limit of normal (ULN; central laboratory) at Screening.
* - Participants with creatinine concentration > 1.5 times the ULN (central laboratory) at Screening.
* - Participants with new onset or worsening or severe cardiac, pulmonary, kidney disease, and liver disease.
* - Participants with malignancies of lymphoid cells such as chronic lymphocytic leukemia, non-Hodgkin's lymphoma, and immunodeficiency with thymoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2026-05-04 (Estimated); Study Completion 2026-05-04 (Estimated)

PRIMARY OUTCOMES:
Trough concentration (Ctrough) Levels of IgPro20 | Up to Week 13
Number of Participants Experiencing Any Treatment-Emergent Adverse Event (TEAEs) or Serious TEAEs | Up to Day 85
Number of TEAEs and Serious TEAEs Events | Up to Day 85
TEAEs and Serious TEAEs Event Rates Per Days with Infusion | Up to Day 85

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (8):
- United States (8):
  - Research Solutions of AZ, Litchfield Park, Arizona
  - Medical Research of Arizona, Scottsdale, Arizona
  - Immunoe Health Centers, Centennial, Colorado
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - Midwest Immunology, Plymouth, Minnesota
  - Washington University, St Louis, Missouri
  - Allergy, Asthma and Clinical Research Center, Oklahoma City, Oklahoma
  - Allergy & Clinical Immunology, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (ie FDA, EMA) is complete and the primary publication is available.
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.